CLINICAL TRIAL: NCT06241690
Title: the Effect of Post-suture Cold Applications on the Pain Level of Children With Sutures
Brief Title: Cold Applications on the Pain Level of Children With Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, DİDEM COŞKUN ŞİMŞEK, Principal Investigator, Firat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: post-suture cold applications
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Child, Only
Keywords: Cold Application; child; Nurse; Pain; suture
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the cold applications in post-suture pain reduces the child's pain (Experimental): The population of the study consists of children aged 12-17 who were treated in the pediatric emergency departments of the designated hospitals between December 2021 and July 2022 and met the working criteria. The sample consists of 300 children who applied to the pediatric emergency service between December 2021 and July 2022 and met the research criteria. Socio-Demographic presentation form and Visual Analog Scale were used as data collection tools. Statistical analysis of the data was made in SPSS 22 package program.
  Interventions: Other: the cold applications in post-suture pain reduces the child's pain

INTERVENTIONS:
Other: the cold applications in post-suture pain reduces the child's pain — The experimental groups was applied cold applications immediately after 20 minutes the suture. Later, The experimental groups was applied cold applications again for 20 minutes 1 hour, 2 hours and 6 hours after the suture.

SUMMARY:
Purpose:This research was conducted as an experimental study with pretest and posttest control groups in order to evaluate the effect of post-suture cold applications on the pain level of children with sutures.

Design and Methods: This study is a randomised controlled study. In the study, there were 150 children in the experimental group and 150 children in the control group.

DETAILED DESCRIPTION:
The experimental groups was applied at the 1st, 2nd and 6th hours after the suture application in the cold applications The different practitioners applied in the Visual Analog Scale after and before in the cold applications to the experimental and control groups

ELIGIBILITY:
Inclusion Criteria:

* parents who agreed to participate in the study

Exclusion Criteria:

* -visually impaired child
* mentally retarded child
* speech impaired children
* without chronic disease

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
this study was measured the effects of cold application in the children after the suture | 1 days
  The experimental groups was applied cold applications immediately after 20 minutes the suture. Later, The experimental groups was applied cold applications again for 20 minutes 1 hour, 2 hours and 6 hours after the suture. The visual Analog Scale were used as data collection tools. The Visual Analog Scale scale was applied before suturing. It was then applied 20 minutes, 1 hour, 2 hours and 6 hours after the suturing procedure.
  The Visual Analog Scale: A minimum of 0 and a maximum of 10 points are obtained from the scale. A high score from the scale indicates a high level of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Elâzığ, Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No